CLINICAL TRIAL: NCT02309736
Title: Device Exposure Registry: A Post-Approval Observational Registry of ReSure Sealant to Track the Incidence of Endophthalmitis After Sealing Corneal Incisions in Patients Undergoing Clear Corneal Cataract Surgery
Brief Title: OTX-14-002: Device Exposure Registry
Status: Withdrawn | Type: Observational
Why Stopped: On going discussions with FDA
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OTX-14-002
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Endophthalmitis
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ReSure Sealant

SUMMARY:
The objective of the study is to collect post-approval data relative to the incidence of endophthalmitis for cataract surgery patients treated with the FDA-approved ReSure Sealant when used by a broad group of physicians under commercial use conditions

ELIGIBILITY:
All patients that receive at least one application of the ReSure Sealant on the operative eye following cataract surgery will be enrolled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of endophthalmitis | Day 30